CLINICAL TRIAL: NCT06373653
Title: Clinical Study of Non-inferiority Between Manzanilla Sophia® and Meticel Ofteno® 0.5% for Providing a Soothing Sensation to the Eyes.
Brief Title: Study of Non-inferiority Between Manzanilla Sophia® and Meticel Ofteno® 0.5% for Providing a Soothing Sensation to the Eyes.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's decision.
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPHMAN-0922/IV
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Eye Strain; Eye Strain of Both Eyes
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Intervention Model Description: Phase IV non-inferiority, open-label, controlled, comparative, multicenter, clinical study.
Masking Description: Open-label,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manzanilla Sophia® (Active Comparator): Matricaria recutita 0.025%, Ophthalmic solution.
  * Dosage: 1 drop every 4 hours (4 daily applications [QID]), during 7 days.
  * Route of administration: Topical ophthalmic.
  Interventions: Drug: Manzanilla Sophia®
- Meticel Ofteno® (Active Comparator): Hypromellose 0.5%. Ophthalmic solution.
  * Dosage: 1 drop every 4 hours (4 daily applications [QID]), during 7 days
  * Route of administration: Topical ophthalmic.
  Interventions: Drug: Meticel Ofteno®

INTERVENTIONS:
Drug: Manzanilla Sophia® — Matricaria recutita 0.025%, Ophthalmic solution.
  Arms: Manzanilla Sophia®
Drug: Meticel Ofteno® — Hypromellose 0.5%, Ophthalmic solution.
  Arms: Meticel Ofteno®

SUMMARY:
This is a phase IV clinical study to demonstrate the non-inferiority of Manzanilla Sophia® compared to Meticel Ofteno® 0.5% in providing restful sensation to the eyes. This will be evaluated by measuring the incidence of unexpected adverse events related to the interventions, the incidence of conjunctival hyperemia and the incidence of sensation of comfort with the application, when applied by the Principal Investigator (PI).

DETAILED DESCRIPTION:
Primary:

-Analog visual eyestrain test score

Secondary:

* Incidence of unexpected adverse events related to the interventions
* Incidence of conjunctival hyperemia
* Incidence of sensation of ocular dryness
* Incidence of ocular irritation
* Incidence of sensation of (sleep-crust)
* Incidence of sensation of comfort with the application, when applied by the Principal Investigator (PI)

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to voluntarily give their signed informed consent.
* Being able to and willing to comply with scheduled visits, treatment plan, and other study procedures.
* Age ≥18 years.
* Women of childbearing potential who have not undergone Bilateral Tubal Occlusion (BTO [Tubal Ligation]), hysterectomy, or bilateral oophorectomy must ensure continuation (initiated ≥ 30 days prior to signing the informed consent form [ICF]) of the use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Present on the analog visual eyestrain test score ≥ 3 on at least 4 of the included questions.

Exclusion Criteria:

* History of hypersensitivity to any of the components of the drugs under investigation.
* Use of contact lenses for a period less than two weeks prior to the start of the study, and during the intervention period of this study.
* In the case of women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Having participated in any clinical research study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* Having a single functional eye.
* Having a history of drug addiction or drug dependence current or within the last two years prior to signing the informed consent.

Elimination Criteria:

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the drugs under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-11 (Estimated); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Analog visual eyestrain test score | Days: 0 (Basal Visit) and 8 (Final Visit).
  The PI will evaluate the analog visual eyestrain test score by applying a direct questionnaire to the subject and allowing the subject to answer it calmly without any pressure.
  The analog visual test score is a questionnaire designed to establish the degree of eyestrain (fatigue) according to its symptomatology. This questionnaire will be as follows for frequency: never (1), sometimes (2), 50% of the time (3), almost all the time (4) and all the time (5).

SECONDARY OUTCOMES:
Incidence of unexpected adverse events related to the interventions | Days 0 (Basal Visit), 3 (Visit 1), 8 (Final Visit) and 10 (Safety Call)
  Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention.
Incidence of conjunctival hyperemia | Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
  Any signs of conjunctival hyperemia in between interventions.
  Conjunctival hyperemia is defined as the red appearance secondary to vasodilatation of the conjunctival blood vessels of variable intensity.
Incidence of sensation of ocular dryness. | Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
  The subject will be questioned directly.
  Ocular dryness is defined as the subjective sensation of dry eye.
Incidence of ocular irritation | Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
  The subject will be questioned directly.
  Ocular irritation is defined as the subjective sensation of eye irritation.
Incidence of sensation of (sleep-crust) | Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
  The subject will be questioned directly.
  Sleep crust is defined as the subjective sensation of the presence of eye discharge.
Incidence of sensation of comfort with the application, when applied by the Principal Investigator (PI) | Day 8 (Final Visit)
  The subject will be questioned directly by de PI during the final visit.

IPD SHARING:
Plan to Share IPD: No